CLINICAL TRIAL: NCT06151314
Title: Bone Density and Marginal Bone Height Changes Around Dental Implants Supporting and Retaining Different Types of Prostheses of Mandibular Kennedy Class VI
Brief Title: Bone Density and Marginal Bone Height Changes Around Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Menatallah Mohamed Elhotieby, researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: National Research Centre
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Implant Site Reaction
Keywords: digital milled partial overdenture; Bone density; Fixed bridge
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "digital milled implant supported removable partial overdenture (Active Comparator): patients received digital milled implant supported removable partial overdenture.
  Interventions: Procedure: Dental implants.
- "implant supported fixed bridge" (Active Comparator): patients received an implant supported fixed bridge
  Interventions: Procedure: Dental implants.

INTERVENTIONS:
Procedure: Dental implants. — 5 conventional implants measuring from 4 to 5 mm in width and 7 to 10mm in length according to the bone width were inserted in the mandible from right premolar area to left premolar area
  Other Names: OXY implants

SUMMARY:
The increased benefits to the edentulous population from implant supported overdenture is overwhelming in terms of better quality of life, emotional stability, improved function, enhanced esthetics and clinical comfort.1-6 Implant supported prosthesis is considered a viable option for partially edentulous patients7. The oral rehabilitation of a long anterior mandibular edentulous span with a fixed or removable implant-supported prosthesis using appropriate prostheses have been a target in oral implant research for the last year. The longevity of any implant prosthesis depends on successful osseointegration and implant stability. Cone beam computed tomography (CBCT ) has also been used extensively for the follow-up of dental implants and is considered one of the tools for assessing implant success

DETAILED DESCRIPTION:
This study will be conducted on 6 patients having mandibula Kennedy Class VI (anterior edentulous span) Each patient will receive 5 dental implants in the interforaminal area. The patients will be randomly categorized into two groups. According to the final restoration they will receive.

Group I: will receive a digital milled implant supported overdenture. While Group II will receive implant supported fixed bridge.

The marginal bone height changes and bone density around the dental implants will be evaluated at the time of prosthesis insertion, after one and three month.

Research Procedures:

1. Patient selection: will be following inclusion and exclusion criteria.
2. 5 implants will be installed in the interforaminal area for each patient.
3. Digital impression, bite registration, try in and delivery of the final prosthesis for each group will follow the conventional methods.
4. The marginal bone height changes and bone density around the dental implants using CBCT will be evaluated at the time of prosthesis insertion, after one and three month.
5. Statistical analysis: Data will be collected, tabulated, and statistically analyzed using Microsoft Excel ® 2016, Statistical Package for Social Science (SPSS)® Ver. 24. and Minitab ® statistical software Ver. 16.

ELIGIBILITY:
Inclusion Criteria:

* non smokers
* Patients having long anterior mandibular edentulous span.
* Highly cooperative and motivated patients.
* Patients Systemically free from any immunosuppressive diseases.
* Patients free from Diabetes, Hypertension, Cancer, any mental or physical diseases.
* Patients not receiving any Radiotherapy or chemotherapy treatment.

Exclusion Criteria:

-Mandibular arch with thin knife edge, flat or flabby ridge, recent extractions, and foreign bodies.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
assessment of change of bone density around dental implants | on the first day,on 1 month ,3months
  bone density was assessed by cone beam computed tomography

SECONDARY OUTCOMES:
assessment of change of bone height around dental implants | on the first day,on 1 month ,3months
  bone height was assessed by cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Menatallah M. Elhotieby, Researcher, Principal Investigator — National Research Centre, Egypt
Locations (2):
- Egypt (2):
  - National Research Centre, Cairo
  - M, Giza